CLINICAL TRIAL: NCT02589834
Title: The Effect of Listening to Quran During Cesarean Section on Postoperative Pain
Brief Title: The Effect of Quran of Post Operative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QPOP
Record Dates: First submitted 2015-10-27; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quran group (Active Comparator): The patients listened to Quran recitation by a compact disc player through an occlusive headphone, started after induction of spinal anesthesia and continued throughout the entire cesarean section duration.
  Interventions: Other: Quran group
- Non-Quran group (No Intervention): Those patients did not listen to Quran and subjected to operative room noise throughout the surgery.

INTERVENTIONS:
Other: Quran group
  Arms: Quran group

SUMMARY:
Postoperative pain management is crucial for surgical patients. Management of postoperative pain entails reducing painful symptoms, improving the quality of recovery and resuming normal daily living activities. In addition to the benefits derived from relieving postoperative pain in women undergoing cesarean section, prolonged immobility as a result of pain during puerperium is associated with risk of thromboembolic disease.

Postoperative pain has negative physiological and psychological impact on patients' well-beings and delays the postoperative recovery. Pain may also impair the mother's ability to provide an optimal care for her infant in the immediate postpartum period. Besides that, it also reduces the maternal ability to breast-feed her infant effectively.

Effective pain relief should not interfere with the mother's ability to move around and care for her infant, and that it results in no adverse neonatal effects in breast-feeding women.

Non-pharmacological techniques for reduction of pain are growing rapidly. Spiritual intervention with listening to Quran recitations as an adjunctive therapy in the postoperative period is a non-pharmacological technique that is inexpensive, non-invasive and has no side-effects. Spiritual and Islamic implication could improve postoperative pain 6-8 hours and 24-30 hours in Muslim patients undergoing abdominal surgery. However, there is limited number of published studies on the effect of spiritual and religious intervention on pain after cesarean section.

Listening to Quran recitation elicits a relaxation response of calmness, mindfulness, and peacefulness in Muslims. Pray therapy results in optimal harmonization, which improves psychological, social, spiritual, and physical health status.

The current study aims to investigate the effects of listening to Quran recitation on pain intensity among patients after cesarean section according to the cultural, social and economic differences in Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Muslim women
* Term (37-40 weeks) gestation
* uncomplicated singleton pregnancy
* scheduled for elective lower segment cesarean section under spinal anesthesia

Exclusion Criteria:

* Any medical diseases
* Hearing impairment
* Any contraindication to spinal anesthesia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Measurement of postoperative pain by Visual analogue scale | 4 months

SECONDARY OUTCOMES:
The amount of postoperative analgesics by mg | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt